CLINICAL TRIAL: NCT01278537
Title: Patient Empowerment and Risk-assessed Treatment to Improve Outcome in the Elderly After Gastrointestinal, Thoracical or Urogenital Cancer Surgery.
Brief Title: Patient Empowerment and Risk-assessed Treatment to Improve Outcome in the Elderly After Onco-surgery
Acronym: PERATECS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Principal Investigator, Claudia Spies, Univ. Prof. Dr. med. Claudia Spies, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PERATECS
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Cancer
Keywords: elderly; cancer surgery; quality of life; empowerment; shared-decision
MeSH Terms: conditions — Neoplasms; Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Empowerment, shared-decision making, (Experimental): Patients receive a booklet with informations. Assessment of health-related risk factors. Assessment of psychological and physical social support Delirium protection. Early mobilization.
  Interventions: Behavioral: Information
- control group (No Intervention)

INTERVENTIONS:
Behavioral: Information — Booklet, motivational interviewing, brief advice
  Arms: Empowerment, shared-decision making,

SUMMARY:
The aims of this study are to investigate whether patient empowerment, including information and decision-aids adapted to the risk and the need of the elderly patient, can improve outcome in an evidence-based modular pathway in terms of

* shortened hospital stay by a reduced postoperative complication rate and
* quality of life in elderly patients compared to control patients receiving standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years and older with abdominal, thoracical or urogenital cancer scheduled for surgery
* Offered patient information and written informed consent
* Confirmed cancer diagnosis via histology
* Mini Mental state > 23
* Life-expectance > 2 months

Exclusion Criteria:

* Participation in another trial according to the German Drug Law 7 days to and 7 days after the operation during the study
* No informed consent
* Emergency patients
* Lacking willingness to save and hand out data within the study
* Accommodation in an institution due to an official or judicial order
* Concurrent malignancies
* Insufficient knowledge of the German language
* In case of the inclusion of a PERATECS - study patient in an adjuvant therapy study during the study period, the patient will be excluded from the PERATECS-study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 690 (Actual)
Dates: Start 2011-02; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | within the first month
Quality of life | within the first year

SECONDARY OUTCOMES:
Readmission rate | within the first three months
Short-term complications | within the first months
Overall mortality | within one year
Depression | within the first year
Stress | within the first month
  Stress induced by postoperative pain, lack of mobilization and PONV.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD Prof., Study Chair — Department of Anesthesiology and Intensive Care Medicine, Campus Virchow-Klinikum and Campus Charité Mitte, Charité - Universitaetsmedizin Berlin
Locations (3):
- Germany (3):
  - Department of Anaesthesiology, Hospital of the Ludwig - Maximilians - University of Munich, München, München
  - Evangelisches Geriatriezentrum Berlin gGmbH, Berlin, State of Berlin
  - Department of Anesthesiology and Intensive Care Medicine, Campus Virchow-Klinikum and Campus Charité Mitte, Charité - Universitaetsmedizin Berlin, Berlin

REFERENCES:
- [Derived] Scholtz K, Borchers F, Morgeli R, Krampe H, Schmidt M, Eckardt-Felmberg R, von Dossow V, Sehouli J, Stief CG, Pohrt A, Spies CD; PERATECS Group. Self-reported exhaustion and a 4-item physical frailty index to predict the incidence of major complications after onco-geriatric surgery. Eur J Surg Oncol. 2024 Jul;50(7):108421. doi: 10.1016/j.ejso.2024.108421. Epub 2024 May 23. PMID 38870573
- [Derived] Mueller A, Spies CD, Eckardt R, Weiss B, Pohrt A, Wernecke KD, Schmidt M; PERATECS-Group. Anticholinergic burden of long-term medication is an independent risk factor for the development of postoperative delirium: A clinical trial. J Clin Anesth. 2020 May;61:109632. doi: 10.1016/j.jclinane.2019.109632. Epub 2019 Oct 24. PMID 31668693
- [Derived] Scholtz K, Spies CD, Morgeli R, Eckardt R, von Dossow V, Braun S, Sehouli J, Bahra M, Stief CG, Wernecke KD, Schmidt M; PERATECS Group. Risk factors for 30-day complications after cancer surgery in geriatric patients: a secondary analysis. Acta Anaesthesiol Scand. 2018 Apr;62(4):451-463. doi: 10.1111/aas.13067. Epub 2018 Jan 22. PMID 29359461
- [Derived] Schmidt M, Eckardt R, Scholtz K, Neuner B, von Dossow-Hanfstingl V, Sehouli J, Stief CG, Wernecke KD, Spies CD; PERATECS Group. Patient Empowerment Improved Perioperative Quality of Care in Cancer Patients Aged >/= 65 Years - A Randomized Controlled Trial. PLoS One. 2015 Sep 17;10(9):e0137824. doi: 10.1371/journal.pone.0137824. eCollection 2015. PMID 26378939